CLINICAL TRIAL: NCT02782130
Title: Epic Allies: A Gaming Mobile Phone Application to Improve Engagement in Care, Antiretroviral Uptake, and Adherence Among Young Men Who Have Sex With Men (YMSM) and Trans Women Who Have Sex With Men
Brief Title: Epic Allies HIV ART Adherence Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 132; 5R44MH102096-03 (NIH)
Record Dates: First submitted 2015-11-10; First posted 2016-05-25 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: HIV
Keywords: HIV; YMSM; Trans women; ART Adherence; Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator): Subjects randomized to the Epic Allies Intervention will download and install the intervention branch of the Epic Allies app and receive a tour of the app guided by site staff. During the 26-week intervention phase, intervention arm subjects will receive daily adherence reminders set up through Epic Allies with tailored feedback for encouragement and reinforcement. Intervention arm subjects will have 24-hour access to all features of Epic Allies and will receive supportive messages from other subjects on the intervention arm.
  Interventions: Behavioral: Epic Allies App Intervention
- Control Group (Placebo Comparator): Subjects randomized to the control arm will download and install the control branch of the Epic Allies app (phone-based notifications only) and be provided with instructions on using the app. During the 26-week intervention phase, the control arm subjects will receive weekly phone-based notifications to encourage the subjects to view educational information presented in the app.
  Interventions: Behavioral: Epic Allies - Control Branch

INTERVENTIONS:
Behavioral: Epic Allies App Intervention — The Epic Allies app addresses barriers to ART adherence through:
  1. Users track health progress through an interactive dashboard, logging daily adherence for those on ART and, optionally, exercise, smoking, alcohol and drug use, and mood. Those not on ART will rate how close they are to getting on it.
  2. Users pick medication reminder timing. The app sends weekly messages to users based on adherence progress and other tracked behaviors.
  3. A key part of the app is contact between users to foster a setting that supports norms for medication-taking, reducing stigma related to HIV status and ART use. Users send and receive encouragement to spur behavior change, recognize positive behaviors, and inspire others to reach an adherence goal.
  4. Users progress through Epic Allies' virtual world, creating allies with other users.
  5. The Daily Dose newspaper has content to improve HIV/ART knowledge, promote disease management and increase drive and self-efficacy.
  Arms: Intervention Group
Behavioral: Epic Allies - Control Branch — Subjects will receive weekly phone-based notifications to encourage the subjects to view educational information presented in the app.
  Arms: Control Group

SUMMARY:
This is a two-arm, randomized-controlled trial (RCT) that will test the acceptability, impact, and long-term sustainability of the Epic Allies intervention application (app), a theory-based mobile app that utilizes game mechanics and social networking features to improve engagement in care, antiretroviral therapy (ART) uptake, ART adherence, and viral suppression among HIV-positive young men who have sex with men (YMSM) and trans women who have sex with men. Subjects will be randomized to either the intervention branch of the Epic Allies app or the control branch of the app.

DETAILED DESCRIPTION:
Implementation of effective interventions for HIV care engagement is necessary to raise the percentage of people living with HIV/Acquired Immunodeficiency Syndrome (AIDS) who are virally suppressed and in continuous care. The ultimate goal of this study is to assess the effectiveness of a mobile phone app that utilizes game mechanics and social networking features to improve engagement in care, and ART uptake and adherence among HIV-positive YMSM and trans women who have sex with men. The high mobile phone ownership among adolescent and young adults supports using intervention tools based in these familiar available technologies. If successful, Epic Allies would be clinically attractive, as adherent patients would require less frequent clinic visits and experience fewer HIV-related secondary infections and financially attractive, as reducing clinic visits and secondary infections. Epic Allies could also greatly impact public health as ART adherence reduces HIV infectivity and subsequently reduces HIV transmission.

This is a two-arm randomized-controlled trial (RCT). All subjects will be randomized either to the intervention arm and receive the Epic Allies intervention branch of the app or to the control arm and receive the phone-based notifications only control branch of the app. Randomization will occur in a 1:1 ratio within each of the two groups (new-to-care and ART-non-adherent) separately, with an equal number of subjects in the intervention and control arms. During the 26-week intervention phase, intervention arm subjects will receive the daily adherence reminders they set up through Epic Allies with tailored feedback for encouragement and reinforcement. Intervention arm subjects will have 24-hour access to all features of Epic Allies. The control arm subjects will receive weekly phone-based notifications to encourage them to view educational information presented in the app. Subjects will attend study visits at Week 13 (during intervention phase), Week 26 (end of intervention phase), and Week 39 (post-intervention phase). In-depth qualitative app satisfaction interviews with a subset of intervention arm subjects will also be conducted to evaluate acceptability of the app and its potential to improve engagement in care, uptake of ART, and ART adherence. Outcome measures will include engagement in care, ART uptake, ART adherence, viral load (VL) change, and VL suppression. The in-depth qualitative app satisfaction interview will assess intervention impact, acceptability, and long-term sustainability.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment, an individual must meet all the criteria listed below.

* Ages 16 years and 0 days through 24 years and 364 days, inclusive, at the time of signed informed consent or assent with parental/legal guardian permission, if applicable;
* Assigned male sex at birth, is of any gender identity, and self-reports a desire to engage or is engaging in sex with men;
* Has documentation of a VL collected within the 12 weeks prior to the Baseline visit that is greater than the LLD for the assay used to test the specimen;
* Be either:

  * New-to-care: Newly entered HIV medical care within the 12 months prior to the Baseline visit; or
  * ART-non-adherent: First entered HIV medical care more than 12 months prior to the Baseline visit;
* Has reliable daily access to an Android- or iOS-based smartphone with a data plan;
* Is able to speak and read English;
* Is willing and able to provide signed informed consent or assent; and
* Parent or legal guardian is willing to provide permission, if applicable.

Exclusion Criteria:

To be considered eligible for enrollment, an individual must not meet any of the criteria listed below.

* Presence of active serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to provide true informed consent/assent or complete the baseline CAPI survey*;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior) at the time of consent/assent or the baseline CAPI survey*;
* Intoxicated or under the influence of alcohol or other substances to such an extent that in the opinion of the study staff, the ability to give true informed/assent is impaired*; or
* At the time of the baseline CAPI survey, intoxicated or under the influence of alcohol or other substances to such an extent that in the opinion of the study staff, the subject's ability to understand and answer the questions may be impaired or negatively impact the integrity of the research data*.

  * NOTE: If consent/assent is obtained prior to enrollment and the Baseline visit date, assessment for these exclusion criteria must be performed again prior to administration of the baseline CAPI survey. If any are present during the Baseline visit, the subject cannot be enrolled; do not administer the CAPI survey. Reassessment of eligibility and enrollment may take place at a later date per the discretion of the treating clinician.

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
VL suppression at 13 weeks | 13 weeks
  VL suppression at 13 weeks is defined as VL below the lower limit of detection (LLD) in the six-week window before the Week 13 visit.
VL suppression at 26 weeks | 26 weeks
  VL suppression at 26 weeks is defined as VL below the lower limit of detection (LLD) in the six-week window before the Week 26 visit.

SECONDARY OUTCOMES:
Self-reported ART adherence | 13 weeks, 26 weeks, and 39 weeks
Retention in HIV Care | 13 weeks, 26 weeks, and 39 weeks
VL suppression at 39 weeks | 39 weeks
  VL suppression at 39 weeks is defined as VL below the lower limit of detection (LLD) in the six-week window before the Week 39 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Hightow-Weidman L, Muessig KE, Egger JR, Vecchio A, Platt A. Epic Allies: A Gamified Mobile App to Improve Engagement in HIV Care and Antiretroviral Adherence among Young Men Who have Sex with Men. AIDS Behav. 2021 Aug;25(8):2599-2617. doi: 10.1007/s10461-021-03222-y. Epub 2021 Mar 19. PMID 33740213
- [Derived] LeGrand S, Muessig KE, Platt A, Soni K, Egger JR, Nwoko N, McNulty T, Hightow-Weidman LB. Epic Allies, a Gamified Mobile Phone App to Improve Engagement in Care, Antiretroviral Uptake, and Adherence Among Young Men Who Have Sex With Men and Young Transgender Women Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 5;7(4):e94. doi: 10.2196/resprot.8811. PMID 29622527